CLINICAL TRIAL: NCT06724575
Title: The EVOLVE Study: A Prospective, Observational Study to Evaluate Patient-centered Outcomes Over 2 Years of Treatment With Tezepelumab in Real-life Clinical Practice in Greece
Brief Title: EVOLVE Study: The Real-life Clinical Practice With Tezepelumab in Greece
Acronym: EVOLVE
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5180R00032
Record Dates: First submitted 2024-11-19; First posted 2024-12-09 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Asthma
Keywords: severe asthma, tezepelumab, real world data, patient reported outcomes, Greece
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tezepelumab is a first-in-class human monoclonal antibody for uncontrolled severe asthma that acts at the top of the inflammatory cascade by targeting thymic stromal lymphopoietin (TSLP), a key epithelial cytokine inducing both Type 2 and non- Type 2 inflammatory pathways. Considering the recent addition of tezepelumab to the severe asthma therapeutic arsenal, there is a need for real-world evidence that can inform treatment-decision making in clinical practice and support regulatory decisions.

EVOLVE is a prospective, observational study designed to generate real-world evidence on patient-reported outcomes of treatment with tezepelumab, assessing the effectiveness over a 2-year period in routine care settings in Greece.

The study plans to enroll 150 adult patients at an allocation ratio of: i) 70 percent Type 2-high/30 percent Type 2-low, and ii) 80 percent biologic naïve/20 percent switching from a prior biologic. Eligible patients must be newly prescribed tezepelumab according to the approved label.

Primary data will be collected at enrollment and 4, 12, 24, 52, 72 and 104 weeks after treatment initiation through visits as per the standard clinical practice in various healthcare settings (20-25 sites) across the country.

The primary objective is to describe the patient-reported asthma symptom control using the Asthma Control Questionnaire (ACQ-6) at baseline and up to 104 weeks post-index. Secondary and exploratory objectives include assessment of quality of life, lung function, exacerbation rate, corticosteroid use, health-care utilization. Novel composite endpoints will also be evaluated such as early clinically important improvement, disease stability, super-response and clinical remission at 2 years, which in the era of precision biologics, have the potential to shift treatment paradigms toward a treat-to-target approach.

Findings of EVOLVE are expected to not only complement evidence obtained from clinical trials, but also to provide valuable insights into the long-term durability of treatment benefits and sustainability of clinical response under pragmatic clinical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged 12 years or older at the time of signing the informed consent/assent form.
* Patients who have been prescribed but not yet initiated treatment with tezepelumab according to the label and local market reimbursement criteria.
* Diagnosis of asthma for at least 52 weeks prior to enrolment date and symptoms confirmed by the Investigator not to be due to alternative diagnoses.
* Receipt of at least one prescription of high-dose Inhaled Corticosteroids (ICS) (according to the Global Initiative for Asthma 2024) during the 52 weeks prior to enrolment date.
* Use of additional asthma maintenance controller medication(s) in addition to ICS either as free- or fixed-drug combination for at least 52 weeks prior to enrolment date.
* Documented history of at least 1 asthma exacerbation during the 52 weeks prior to enrolment date.
* Asthma Control Questionnaire (ACQ-6) score ≥1.5 (indicating inadequate asthma symptom control) at enrolment.
* Availability of at least one Blood Eosinophil Count (BEC) measurement (in medical records) in the 52-week period prior to enrolment date.
* Availability of participants' medical records for asthma exacerbations and unscheduled Health Care Resource Utilization (HCRU) for the 52 weeks prior to enrolment date.
* Patients are able to understand and complete the Patient-Reported Outcome (PROs).
* Provision of signed and dated written informed consent/assent (as applicable).

Exclusion Criteria:

* Any contraindication to tezepelumab as per the approved product label or in the opinion of the Investigator.
* Concurrent or recent (<30 days before the index date) treatment with biologics for asthma, with the exception of stable allergen immunotherapy (defined as a stable dose and regimen at the time of enrolment).
* Participation in an observational study that might, in the Investigator's opinion, influence the assessment for the current study, or participation in an interventional clinical trial in the last 3 months.
* Currently pregnant (or intention to become pregnant) or lactating women.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population from private practices and hospital clinics specializing in the management of Severe Asthma, in geographically diverse locations throughout Greece, with a balanced representation of public, academic and private sector in Greece.
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2024-12-17 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the ACQ-6 score at baseline and up to 104 weeks post-index | Before treatment initiation and at Weeks 4, 12, 24, 52, 72, 104 after treatment initiation
  Asthma Control Questionnaire-6 (ACQ-6) score at different timepoints Change in ACQ-6 score from baseline Proportion of patients with ACQ-6 response (i.e., achieving the Minimum Clinically Important Difference (MCID) of ≥0.5 reduction in score from baseline) Proportion of patients with major improvement in asthma control (defined as decrease in ACQ-6 score ≥1 point [i.e., 2xMCID] from baseline) Proportion of patients with well-controlled asthma (ACQ-6 score ≤ 0.75) Proportion of patients with ACQ-6 score in categories 0.75 to <1.5 and ≥1.5 Time to ACQ-6 score response

SECONDARY OUTCOMES:
Change in asthma-specific HRQoL using the SGRQ at baseline and up to 52 weeks post-index | Before treatment initiation and at Weeks 24 and 52 after treatment initiation
  St. George's Respiratory Questionnaire (SGRQ) total and component scores at different timepoints Change in SGRQ total and component scores from baseline Proportion of patients with SGRQ response (≥4-point reduction in total score from baseline)
Change in FEV1 (forced expiratory volume in 1 second) at baseline and up to 104 weeks post-index | Before treatment initiation and at Weeks 4, 12, 24, 52, 72 and 104 after treatment initiation
  To describe the pre- and post-BD (Bronchodilation) FEV1, as well as the changes from baseline in pre- and post-BD FEV1 in patients receiving Tezepelumab.
Change in FVC (Forced Vital Capacity) at baseline and up to 104 weeks post-index | Before treatment initiation and at Weeks 4, 12, 24, 52, 72 and 104 after treatment initiation
  To describe the pre- and post-BD (Bronchodilation) FVC, as well as the changes from baseline in pre- and post-BD FVC in patients receiving Tezepelumab.
Change in pre-BD FEF25-75 (Forced Expiratory Flow) at baseline and up to 104 weeks post-index | Before treatment initiation and at Weeks 4, 12, 24, 52, 72 and 104 after treatment initiation
  To assess the pre-BD (Bronchodilation) FEF25-75, as well as the changes from baseline in pre-BD FEF25-75 in patients receiving Tezepelumab
Change in lung function at baseline and up to 104 weeks post-index | Before treatment initiation and at Weeks 4, 12, 24, 52, 72 and 104 after treatment initiation
  To evaluate the proportion of pre- and post-BD (Bronchodilation) FEV1 responders (≥5 percent or ≥100 mL improvement from baseline)
Change in asthma exacerbations in the 52 and 104 weeks post-index | During 52 weeks before treatment initiation and 52 and 104 weeks after treatment initiation
  To describe (a) Annualised Asthma Exacerbation Rate (AAER), (b) change in AAER from the 52 week period pre-index to the 52- and 104- week period post-index and (c) change in AAER associated with hospitalization or ED visit from the 52 week period pre-index to the 52- and 104- week period post-index
Proportion of patients with asthma exacerbations in the 52 and 104 weeks post-index | During 52 weeks before treatment initiation and 52 and 104 weeks after treatment initiation
  To assess the (a) proportion of patients with asthma exacerbations after 52 and 104 weeks of treatment with Tezepelumab, (b) the proportion of patients who completed the 52 week period post-index with any reduction, ≥50 percent, and 100 percent reduction in total number of asthma exacerbations compared with baseline period, and (c) the proportion of patients with asthma exacerbations resulting in hospitalization, and number of hospital days owing to exacerbations (total and averaged per patient) in the 52 week periods pre- and post-index
Time to first asthma exacerbation from index date | Until 104 weeks after treatment initiation
  To describe the time to first asthma exacerbation from index date of treatment with Tezepelumab
Proportion of patients with asthma-related Systemic Corticosteroids (SCS) and Inhaled Corticosteroids (ICS) use during the 52 week-period pre- and post-index | During 52 weeks before treatment initiation and 52 weeks after treatment initiation
  To assess (a) the proportion of patients with any SCS or ICS use, (b) the proportion of patients who completed the 52 week period post-index with any reduction, ≥25 percent, ≥50 percent ≥75 percent and 100 percent reduction in SCS cumulative dose (in prednisone equivalent dose) compared with baseline period, (c) the proportion of patients who completed the 52 week period post-index with any reduction, ≥50 percent (medium dose) and ≥75 percent (low dose) reduction in ICS dose compared with baseline period, (d) the proportion of patients requiring long-term (>30 consecutive days) SCS use, and the proportion of patients requiring long-term (>30 consecutive days) ICS use.
Change in asthma-related Systemic Corticosteroids (SCS) and Inhaled Corticosteroids (ICS) use during the 52 week-period pre- and post-index | During 52 weeks before treatment initiation and 52 weeks after treatment initiation
  To evaluate the change in cumulative annualized SCS and ICS dose through the 52 week periods pre- and post-index
Time to earliest Systemic Corticosteroids (SCS) use from index date | During 52 weeks before treatment initiation and 52 weeks after treatment initiation
  To describe the time to earliest SCS use from index date among patients that used SCS
Change in rate and duration of asthma-related HCRU for the 52 weeks pre- and post-index | During 52 weeks before treatment initiation and during 52 and 104 weeks after treatment initiation
  Number and proportion of patients with any asthma-related Healthcare Resource Utilization (HCRU) and type of HCRU [i.e., hospitalisations/ Emergency Department (ED) visits (without hospitalisation)/unscheduled outpatient or physician visits] Annualized rate of (a) asthma-related visits leading to hospitalisation, (b) ED visits (without hospitalisation), and (c) unscheduled outpatient or physician visits Duration (total and Intensive Care Unit Length of Stay) of asthma-related hospitalisations
Changes in proportion of participants achieving (a) asthma disease stability or (b) partial stability up to 104 weeks post-index | At weeks 4, 12, 24, 52, 72 and 104 after treatment initiation
  To evaluate (a) the proportion of participants achieving stable disease [all 4 criteria are met: i) Asthma Control Questionnaire-6 (ACQ-6) < 1.5 at post-index timepoint; ii) pre-bronchodilator forced expiratory volume in one second (Pre-BD FEV1) at post-index timepoint/pre-BD FEV1 at baseline >0.95; iii) ≥50 percent reduction in the annualized number of exacerbations in the follow-up period; iv) ≥ 50 percent reduction in oral corticosteroid (OCS) use in the follow-up period], and (b) the proportion of participants with partial disease stability (1 criterion, 2 criteria, and 3 criteria are met)
Duration of therapy at 52 and 104 weeks post-index | At Week 52 and 104 after treatment initiation or at the moment of treatment discontinuation through study completion, an average of 2 years (104 weeks)
  To assess the duration of treatment with tezepelumab, as well as the time to tezepelumab treatment discontinuation
Discontinuation rate at 52 and 104 weeks post-index | At Week 52 and 104 after treatment initiation or at the moment of treatment discontinuation through study completion, an average of 2 years (104 weeks)
  To evaluate (a) the rate of for tezepelumab treatment discontinuation and (b) the proportion of participants switching to other biologics for asthma. To describe also the reasons for tezepelumab treatment discontinuation, using a pre-defined checklist.

CONTACTS AND LOCATIONS:
Locations (8):
- Greece (8):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Corfu
  - Research Site, Crete
  - Research Site, Ioannina
  - Research Site, Larissa
  - Research Site, Pátrai
  - Research Site, Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home